CLINICAL TRIAL: NCT00192400
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial to Compare the Safety, Tolerability, Immunogenicity and Efficacy of One Dose and Two Doses of a Liquid Formulation of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T) Compared With Placebo in Healthy Children
Brief Title: Trial to Assess the Safety and Tolerability of the Liquid Formulation of CAIV-T in Healthy Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: D153-P504
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Healthy
MeSH Terms: interventions — FluMist

INTERVENTIONS:
Biological: CAIV-T

SUMMARY:
The purpose of this study is to determine the efficacy of the liquid formulation of CAIV-T against culture confirmed influenza illness in healthy children aged at least 6 months and less than 36 months.

ELIGIBILITY:
Inclusion Criteria: (First Season)

* who is aged at least 6 months and less than 36 months of age at the time of enrollment;
* who is in good health as determined by medical history, physical examination and clinical judgement;
* whose parent(s)/legal guardian(s) have provided written informed consent after the nature of the study has been explained;
* who, along with their parent(s)/legal guardian(s), will be available until the completion of the first season's surveillance phase;
* whose parent(s)/legal guardian(s), can be reached by study staff for the post-vaccination contacts [telephone, clinic or home visit].

(Second Season)

* who was enrolled into the first season of the trial and received at least one vaccination in the primary series;
* who completed the safety and efficacy evaluations during the first season surveillance phase;
* who is in good health as determined by medical history, physical examination and clinical judgement;
* whose parent(s)/legal guardian(s) have provided written informed consent for the second season of the trial after the nature of the study has been explained;
* who, along with their parent(s)/legal guardian(s), will be available until the completion of the second season's surveillance phase;
* whose parent(s)/legal guardian(s), can be reached by study staff for the post-vaccination contacts [telephone, clinic or home visit].

Exclusion Criteria: (First Season)

* whose parent(s)/legal guardian(s) are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* have an immunosuppressed or an immunocompromised individual living in the same household;
* who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational);
* who, in the two weeks prior to entry into this study, received a dose of any influenza treatment (commercial or investigational);
* with a documented history of hypersensitivity to egg or egg protein or any other component of the assigned study vaccine;
* with a clinically confirmed respiratory illness with wheezing within two weeks prior to enrollment;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrollment or for which use is anticipated during the study;
* who were administered any live virus vaccine within one month prior to enrollment or expected to receive another live virus vaccine within one month of vaccination in this study;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results.

If any of these criteria are met following enrolment, the subject will be excluded from subsequent vaccine dosing.

Note: Pregnancy in a household member or any person who has regular contact with the subject is not a contraindication to the enrollment or ongoing participation of the subject in the study.

(Second Season)

* whose parent(s)/legal guardian(s) are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroid of a dose equivalent to 2 mg/kg/day or greater of prednisolone or equivalent to a total of 20 mg/day or greater for children who weigh more than 10 kg, for more than 14 days duration until 2 weeks after corticosteroids have been discontinued;
* who received any blood products, including immunoglobulin, in the period from six months prior to the second season vaccination through to the conclusion of the study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to the second season vaccination through to the conclusion of the study;
* have an immunosuppressed or an immunocompromised individual living in the same household;
* who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational) with the exception of the primary series of study vaccine (CAIV-T/placebo);
* who, in the two weeks prior to receiving the second season vaccination, received a dose of any influenza treatment (commercial or investigational);
* with a documented history of hypersensitivity to egg or egg protein or any other component of the assigned study vaccine (CAIV-T/placebo);
* with a clinically confirmed respiratory illness with wheezing within two weeks prior to receiving the second season vaccination;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to receiving the second season vaccination or for which use is anticipated during the study;
* who were administered any live virus vaccine within one month prior to receiving the second season vaccination or expected to receive another live virus vaccine within one month of receiving the second season vaccination;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results.

Note: Pregnancy in a household member or any person who has regular contact with the subject is not a contraindication to the enrollment or ongoing participation of the subject in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2160
Dates: Start 2002-03; Study Completion 2002-11

PRIMARY OUTCOMES:
The primary endpoint for efficacy is the first episode in the first season in a study child of a culture-confirmed influenza illness, caused by community-acquired subtypes antigenically similar to those contained in the vaccine.

SECONDARY OUTCOMES:
The first episode in the second season in a study child of a culture-confirmed influenza illness, caused by community-acquired subtypes antigenically similar to those contained in the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC

REFERENCES:
- [Derived] Bracco Neto H, Farhat CK, Tregnaghi MW, Madhi SA, Razmpour A, Palladino G, Small MG, Gruber WC, Forrest BD; D153-P504 LAIV Study Group. Efficacy and safety of 1 and 2 doses of live attenuated influenza vaccine in vaccine-naive children. Pediatr Infect Dis J. 2009 May;28(5):365-71. doi: 10.1097/INF.0b013e31819219b8. PMID 19395948